CLINICAL TRIAL: NCT03671590
Title: A Phase 1 Pharmacokinetic and Pharmacodynamic Study of TG-1701, an Irreversible Bruton's Tyrosine Kinase Inhibitor, in Patients With B-Cell Malignancies
Brief Title: Study of TG-1701, an Irreversible Bruton's Tyrosine Kinase Inhibitor, in Patients With B-Cell Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-1701-101
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — umbralisib; ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: TG-1701 Monotherapy (Experimental): Participants will receive TG-1701 oral daily dose. As per protocol v6.0, participants from this arm will be transitioned to the long-term extension arm to receive TG-1701 monotherapy.
  Interventions: Drug: TG-1701
- Arm 2: TG-1701 + Ublituximab + Umbralisib (Experimental): Participants will receive TG-1701, oral dose in combination with ublituximab, oral dose and umbralisib, fixed IV infusion on specific Days of Cycles 1 and 2, followed by maintenance infusions in Cycles 3 to 6 (Cycle=28 days). As per protocol v6.0, participants from this arm will be transitioned to the long-term extension arm to receive TG-1701 monotherapy.
  Interventions: Drug: TG-1701; Drug: Umbralisib; Biological: Ublituximab
- Arm 3: Long Term Safety Extension - TG-1701 Monotherapy (Experimental): All the ongoing participants from Arm 1 and 2, will be transitioned to TG-1701 monotherapy in long-term extension period, per protocol version 6.0.
  Interventions: Drug: TG-1701

INTERVENTIONS:
Drug: TG-1701 — Oral daily dose
Drug: Umbralisib — Oral Daily Dose
  Other Names: TGR-1202
  Arms: Arm 2: TG-1701 + Ublituximab + Umbralisib
Biological: Ublituximab — IV infusion
  Other Names: TG-1101
  Arms: Arm 2: TG-1701 + Ublituximab + Umbralisib

SUMMARY:
This is a Phase 1 trial to evaluate the safety, pharmacokinetics and efficacy of TG-1701, a Bruton's Tyrosine Kinase (BTK) inhibitor in patients with relapsed or refractory B-cell malignancies.

DETAILED DESCRIPTION:
This Phase I clinical trial aims to evaluate the safety of the investigational drug TG-1701 both as a single-agent and in combination with other investigational drugs, specifically ublituximab and umbralisib. As per protocol v6.0, combination therapy (TG-1701 + Ublituximab + Umbralisib) will be discontinued and the participants from Arm 1 and 2 will be transitioned to the long-term extension period to receive TG-1701 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory histologically confirmed B-cell lymphoma or CLL
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2
* Adequate organ function

Exclusion Criteria:

* Prior therapy with a BTK inhibitor (ibrutinib, acalabrutinib, other)
* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Known hepatitis B virus, hepatitis C virus or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose acceptable for participants | From first dose up to 30 days post last dose (Up to approximately 4.8 years)
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities.

SECONDARY OUTCOMES:
Overall Response Rate | Up to approximately 4.8 years
  To assess the overall response rate (ORR) in patients with hematologic malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Constantine S. Tam, MD, Study Chair — St. Vincents Hospital
Locations (8):
- Australia (4):
  - TG Therapeutics Investigational Trial Site, East Melbourne, Victoria
  - TG Therapeutics Investigational Trial Site, Fitzroy, Victoria
  - TG Therapeutics Investigational Trial Site, Nedlands, Western Australia
  - TG Therapeutics Investigational Trial Site, Adelaide
- Poland (4):
  - TG Therapeutics Investigational Trial Site, Krakow
  - TG Therapeutics Investigational Trial Site, Lublin
  - TG Therapeutics Investigational Trial Site, Warsaw
  - TG Therapeutics Investigational Trial Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No